CLINICAL TRIAL: NCT04648865
Title: A Single-Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of LY3537031 in Healthy Participants
Brief Title: A Study of LY3537031 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17756; J2S-MC-GZMA (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06-15

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3537031 (Experimental): LY3537031 administered subcutaneously (SC).
  Interventions: Drug: LY3537031
- Placebo (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3537031 — Administered SC.
  Arms: LY3537031
Drug: Placebo — Administered SC.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3537031 in healthy participants. The blood tests will be performed to check how much LY3537031 gets into the bloodstream, how long the body takes to eliminate it and how body handles LY3537031. Each participant will receive a single dose of LY3537031 or placebo. The study will last up to approximately 71 days for each participant, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female not of childbearing potential
* Have a body mass index (BMI) between 19 and 35 kilograms per square meter (kg/m²) and a body weight ≥ 54 kilograms (kg)
* Have blood pressure, pulse rate, blood and urine laboratory test results that are acceptable for the study
* Have veins suitable for blood sampling

Exclusion Criteria:

* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Have a diagnosis or history of cancer or malignant disease within 5 years
* Have been treated with prescription and over-the-counter medications that promote weight loss within 3 months prior to screening
* Show clinical evidence of syphilis, HIV, hepatitis C, or hepatitis B, and/or test positive
* Have undergone any form of bariatric surgery
* Have previously completed or withdrawn from this study
* Are currently participating in or completed a clinical trial within the last 3 months
* Regularly use known drugs of abuse or with positive drug results
* Smoke >10 cigarettes per day or the equivalent, or are unable or unwilling to refrain from nicotine during CRU admission

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through final follow-up at approximately Day 43
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3537031 | Baseline through final follow-up at approximately Day 43
  PK: AUC of LY3537031
PK: Maximum Concentration (Cmax) of LY3537031 | Baseline through final follow-up at approximately Day 43
  PK: Cmax of LY3537031

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Clinical Research Hospital Tokyo, Shinjuku-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No